CLINICAL TRIAL: NCT02110498
Title: Early Detection of Pancreatic Cystic Neoplasms
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Lustgarten Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00084662
Record Dates: First submitted 2014-03-30; First posted 2014-04-10 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Cysts; Intraductal Papillary Mucinous Neoplasm; Pancreatic Mucinous-Cystic Neoplasm; Cystic, Mucinous and/or Serous Neoplasm; Solid Pseudopapillary Tumour of the Pancreas
Keywords: Pancreatic cyst; IPMN; SCA; SPN; MCN; pancreatic cystic neoplasm
MeSH Terms: conditions — Pancreatic Cyst

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pancreatic cyst fluid, blood
Oversight: Data Monitoring Committee: No

SUMMARY:
This research is being done to learn more about pancreatic cysts. The tests that are currently available are imperfect at determining exactly what type of pancreatic cyst a person has, which cysts contain cancer, or what the risk is of developing cancer in the future. The aim of this study is to use a combination of clinical, imaging, cyst fluid analysis, and molecular markers to try to help develop better tools to answer these questions.

DETAILED DESCRIPTION:
Incidental pancreatic cysts are increasingly recognized due to the widespread use of cross-sectional imaging techniques such as CT and MRI. A number of lesions in the pancreas can form cysts, including serous cystadenomas (SCA), mucinous cystic neoplasms (MCNs), intraductal papillary mucinous neoplasms (IPMNs), solid-pseudopapillary neoplasms (SPNs), and pseudocysts. SCAs and pseudocysts are considered benign; whereas SPNs are considered malignant and require surgical resection. IPMNs and MCNs are considered neoplasms with malignant potential, although the exact risk of malignant progression of these cysts is unknown. Currently, MCN are all surgically resected, whereas IPMN are resected if they have features suspicious for malignancy.

However, current diagnostic tests cannot always reliably distinguish harmless from potentially harmful cysts. Recent studies conducted at Johns Hopkins have shown that each cyst type has unique genetic features that could be used as diagnostic biomarkers. In this study, clinical, imaging data and cyst fluid analysis of individuals with pancreatic cysts will be collected. In patients who undergo an endoscopic ultrasound (EUS) procedure, if a fine needle aspiration (EUS-FNA) is performed, and there is extra cyst fluid left after standard clinical tests have been sent, the extra cyst fluid will be submitted for molecular marker analysis. If an individual undergoes surgery to remove the cyst, cyst fluid will be collected after the cyst has been removed. In addition, a small amount of blood will be collected at the time of the EUS or surgical procedure.

AIMS: The general aim is to propose and prospectively validate a diagnostic approach and model for prediction of mucinous versus non-mucinous, and malignant versus non-malignant, pancreatic cysts using a combination of clinical, radiologic, and biomarker characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age 18 years and older with pancreatic cyst.

Exclusion Criteria:

* Individuals with ASA class 4 or greater.
* Inability to provide informed consent.
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any individual with a pancreatic cyst seen at the Johns Hopkins Hospital or other participating Institutions.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2014-03; Primary Completion 2025-03 (Actual); Study Completion 2025-03 (Actual)

PRIMARY OUTCOMES:
To develop and prospectively validate a panel of molecular markers to differentiate benign pancreatic cysts from those with malignant potential using surgical pathology as the gold standard | 3 years

SECONDARY OUTCOMES:
To determine the sensitivity, specificity, and overall accuracy of imaging (CT, MRI and EUS) in patients with pancreatic cysts | 3 years
  Sensitivity and specificity of imaging results in identifying malignant and mucinous cysts will be calculated using the pathology result as the reference gold standard. The overall accuracy of the imaging results, defined as percent agreement with pathology, will also be calculated. Estimates will be reported with exact binomial 95% confidence intervals.

OTHER OUTCOMES:
To determine the proportion of patients with malignancy in operable pancreatic cysts | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marie O'Broin-Lennon, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States